CLINICAL TRIAL: NCT06400290
Title: Multivessel Balloon Occlusion to Investigate Obstructive Coronary Artery Disease and aNgina
Acronym: ORBITA-MOON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government); Mid and South Essex NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); St George's Healthcare NHS Trust (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21HH7372; NIHR302493 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2024-04-24; First posted 2024-05-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Stable Angina; Multivessel Coronary Artery Disease
Keywords: Angina; Multi-vessel coronary artery disease; Symptoms; Placebo-controlled symptom assessment
MeSH Terms: conditions — Angina, Stable; Angina Pectoris | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: All participants will partake in the same research protocol.
Masking Description: Participants and outcomes assessors will be briefly blinded during the experimental research procedure, during the placebo-controlled balloon inflations when they are asked to report their symptoms. Once the inflations have been completed, all patients will go on to have stents and the blinded part of the protocol will be over.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with stable angina (Experimental): Patients who:
  1. Are symptomatic with angina
  2. Have anatomically severe multi-vessel coronary artery disease
  3. Have physiological evidence of myocardial ischaemia
  Interventions: Procedure: Percutaneous coronary intervention (PCI); Diagnostic Test: Symptom assessment during experimentally induced ischaemia

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Coronary artery stenting for stable angina
Diagnostic Test: Symptom assessment during experimentally induced ischaemia — Transient experimental balloon occlusion across coronary stenosis to determine the symptoms conferred by ischaemia at this stenosis.

SUMMARY:
ORBITA-MOON is a double-blinded, placebo-controlled experimental study that aims to understand how the different coronary artery stenoses contribute to overall clinical angina in patients with multi-vessel coronary artery disease. This study will investigate the symptoms conferred by each stenosis, induced by experimental ischaemia, for 60 patients with multi-vessel coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for PCI due to angina
* Anatomical evidence of significant multi-vessel coronary stenosis defined by either:

  1. ≥70% stenosis in two or more coronary arteries of ≥2.5mm visual diameter stenosis, on invasive coronary angiography (ICA)
  2. Severe stenosis in ≥2 coronary arteries of ≥ 2.5mm visual diameter stenosis, on CTCA
* Physiological evidence of ischaemia with a positive test corresponding to the coronary arteries to be stented, on at least one of the following:

  * dobutamine stress echocardiogram
  * cardiac MRI
  * myocardial perfusion study
  * invasive metrics of coronary physiology

Exclusion Criteria:

* Recent acute coronary syndrome
* Previous coronary artery by-pass graft surgery (CABG)
* Significant left main stem disease
* Chronic total occlusion in the target artery(s)
* Moderate to severe valvular disease
* Moderate to severe left ventricular impairment
* Contraindication to PCI or a drug-eluting stents
* Contraindication to antiplatelet therapy
* Contraindication to adenosine
* Pregnant
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Placebo-controlled similarity score during induced ischaemia at the coronary stenosis | Intra-procedural
  The patient scores the similarity of the angina experienced during the experimental balloon inflation procedure against the angina experienced before the procedure between 0-10 (Higher Score = Most similar)

SECONDARY OUTCOMES:
Placebo-controlled intensity score during induced ischaemia at the coronary stenosis | Intra-procedural
  The patient scores the severity of the angina experienced during the experimental balloon inflation procedure between 0-10 (Higher Score = More severe)
Angina symptom type during induced ischaemia at the coronary stenosis | Intra-procedural
  The patient will list all symptoms experienced during the experimental balloon inflation procedure.
Change in angina symptom score | 57 days
  Fractional Change in Angina Frequency (0-1) (Lower Score = Better Outcome)
Angina severity as assessed by Canadian Cardiovascular Society Class | 57 days
  Canadian Cardiovascular Society Class (0-IV) (Lower Score = Better Outcome)
Angina severity as assessed by MRC dyspnoea scale | 57 days
  MRC dyspnoea score (1-5) (Lower Score = Better Outcome)
Physical limitation, angina stability, quality of life, angina frequency, freedom from angina as assessed with the Seattle Angina Questionnaire | 57 days
  Seattle Angina Questionnaire (0-100), (Higher Score = Better Outcome)
Quality of Life assessed with the EQ-5D-5L questionnaire | 57 days
  EQ-5D-5L Questionnaire (-0.59 to 1), (Higher Score = Better Outcome)
Psychological impact of angina as assessed by the PHQ-9 questionnaire | 57 days
  PHQ-9 Questionnaire (0-27), (Lower Score = Better Outcome)
Psychological impact of angina as assessed by the Beck Depression Inventory | 57 days
  Beck Depression Inventory (0-63), (Lower Score = Better Outcome)
Psychological impact of angina as assessed by the Coping Strategies Questionnaire | 57 days
  Coping Strategies Questionnaire (13-52), (Higher Score = Better Outcome)
Psychological impact of angina as assessed by the Pain Catastrophizing Scale | 57 days
  Pain Catastrophizing Scale (0-52), (Lower Score = Better Outcome)
Psychological impact of angina as assessed by the Profile of mood states questionnaire | 57 days
  Profile of mood states Questionnaire (0-44), (Lower Score = Better Outcome)
Psychological impact of angina as assessed by the SCL-90 Questionnaire | 57 days
  SCL-90 Questionnaire (0-360), (Lower Score = Better Outcome)
Need for anti-anginal medication introduction and uptitration | 57 days
  Has the patient required anti-anginal introduction and/or uptitration. (Score 0-1), (0 = no, 1 = yes)
Angina type as assessed by the Rose Chest Pain Questionnaire | 57 days
  Rose Chest Pain Questionnaire (Score positive or negative), (Positive = pain suggestive of coronary heart disease, negative = pain not suggestive of coronary artery disease)
Angina type as assessed by the McGill Pain Questionnaire | 57 days
  McGill Pain Questionnaire (Score 0-78), (Lower Score = Better Outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Al-Lamee, PhD MRCP, Principal Investigator — Imperial College London
Locations (9):
- United Kingdom (9):
  - Essex Cardiothoracic Centre, Basildon
  - Royal Bournemouth Hospital, Bournemouth
  - Royal Sussex County Hospital, Brighton
  - Imperial College NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - St Georges University Hospital, London
  - Nottingham City Hospital, Nottingham
  - Portsmouth Hospitals University NHS Trust, Portsmouth
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No